CLINICAL TRIAL: NCT02837978
Title: Prospective Clinical Study to Observe the Efficacy and Safety of Tacrolimus in Refractory Rheumatoid Arthritis Patients for 6 Months Treatment in China
Brief Title: The Efficacy and Safety of Tacrolimus in Refractory Rheumatoid Arthritis Patients for 6 Months and Long-term Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Qiang Shu (Other)
Responsible Party: Sponsor-Investigator, Qiang Shu, Chief Physician, Qilu Hospital of Shandong University
Organization: Qilu Hospital of Shandong University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tacrolimus RA QiluH
Record Dates: First submitted 2016-07-13; First posted 2016-07-20 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Arthritis, Rheumatoid
Keywords: Arthritis, Rheumatoid; Tacrolimus; Treatment outcome; Safety
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Tacrolimus; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tacrolimus group (Experimental): RA patients treated with tacrolimus, without MTX
  Interventions: Drug: Tacrolimus
- Tacrolimus + MTX group (Active Comparator): RA patients treated with tacrolimus and MTX
  Interventions: Drug: Tacrolimus; Drug: MTX

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus capsule: 0.5mg to 1mg, po, twice per day (Bid)，adjusted by its concentration in blood or due to patient response. Then may titer down until the endpoint.
  Other Names: FK506
Drug: MTX — MTX：5mg to 15mg, po, once per week (Qw) until the endpoint or adjusted due to unacceptable toxicity develops.
  Other Names: methotrexate
  Arms: Tacrolimus + MTX group

SUMMARY:
This study is designed to observed prospectively the efficacy and safety of 6 months and long-term treatment of Tacrolimus alone or with methotrexate (MTX) in moderate and severe Chinese RA patients who shown insufficiency response or intolerance to DMARDs

DETAILED DESCRIPTION:
This study will enroll 150 cases of refractory rheumatoid arthritis (RA) patients in Chinese，who are in moderate or severe disease activity and insufficiency response or intolerance to DMARDs. The participants plan to be treated with Tacrolimus alone, or along with methotrexate (MTX) if participants were tolerant to MTX. The efficacy and safety of 6 month Tacrolimus treatment in RA patients will be evaluated with DAS28 and other disease activity indices.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed based on 1987 ACR classification criteria for rheumatoid arthritis;
2. Age ≥18 years;
3. Patients have a history of DMARDs including csDMARDs（methotrexate，leflunomide, hydroxychloroquine, iguratimod, sulfasalazine) or any biologic DMARDs（TNFi，tocilizumab or Tofacitinib），prednisone or Chinese traditional Medicine（tripterygium Glycosides，Sinomenine）for 3 months, but couldn't achieve clinical remission， or couldn't tolerate one or more DMARDs;
4. Medium or high disease activity (DAS28≥3.2);
5. Extra-articular manifestations (such as pulmonary fibrosis, proteinuria, leukopenia and peripheral neuropathy ) of RA patients are stable or no significant progress;
6. Dose of prednisone and NSAIDs remain stable for at least one month.

Exclusion Criteria:

1. Patients with acute or chronic infections such as active bacterial, viral, fungal, tuberculosis infection or active hepatitis B;
2. Platelet counts(PLT) <80 x 10^9 / L, or white blood cell (WBC) <3 x 10^9 / L;
3. Propionate acid aminotransferase (ALT) or aspartate aminotransferase (AST) is two times higher than the upper limit of normal;
4. Renal insufficiency: serum Cr ≥ 176 umol / L;
5. Pregnant or nursing women (breastfeeding) ；
6. Patients has a history of malignancy (cure time in less than 5 years);
7. Patients with severe or poorly controlled hypertension, diabetes or cardiac dysfunction;
8. Other comorbidities that cannot be treated with immune suppressants. In addition, once patients experience severe adverse drug reactions、ineffective treatment or rapid progression of rheumatoid arthritis, then quit this research.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline Disease Activity Score 28 (DAS28-ESR) at 24 and longer weeks. | 12 week, 24week,36 week,48 week,72 week,96 week,120 week,144 week
  Change from baseline Disease Activity Score 28 (DAS28) erythrocyte sedimentation rate (ESR) at 24 and longer weeks.

SECONDARY OUTCOMES:
Change from baseline ACR20 response rate at 24 and longer weeks. | 12 week, 24week,36 week,48 week,72 week,96 week,120 week,144 week
  Change from baseline ACR20 response rate at 24 and longer weeks.
The clinical remission rate at 24 and longer weeks. | 12 week, 24week,36 week,48 week,72 week,96 week,120 week,144 week
  The percentage of patients who achieve clinical remission patients at the endpoint or withdraw timepoint.
  High disease activity: DAS28 score exceeding 5.1, Moderate disease activity: DAS28 score of exceeding 3.2 to 5.1, Low disease activity (LDA): DAS28 score of less than or equal to 3.2, Remission: DAS28 score is less than 2.6. clinical remission means Low disease activity or remission.
Clinical response was analyzed using the European League Against Rheumatism (EULAR) improvement criteria. | 12 week,3 week, 24week,36 week,48 week,72 week,96 week,120 week,144 week
  Good response: ΔDAS28 > 1.2 and DAS28 ≤3.2； Moderate response: 1.2 ≥ΔDAS28 > 0.6 and 3.2<DAS28 ≤5.1； or ΔDAS28 > 1.2 and still DAS28>3.2； No response:ΔDAS28≤0.6； or 1.2≥ΔDAS28 > 0.6 and DAS28>5.1。
Change from baseline Simplified Disease Activity Index (SDAI) at 24 and longer weeks. | 12 week, 24week,36 week,48 week,72 week,96 week,120 week,144 week
  Change from baseline Simplified Disease Activity Index (SDAI) at 24 and longer weeks.
Change from baseline Clinical disease activity index (CDAI) at 24 and longer weeks. | 12 week, 24week,36 week,48 week,72 week,96 week,120 week,144 week
  Change from baseline Clinical disease activity index (CDAI) at 24 and longer weeks.
Change from baseline Erythrocyte Sedimentation Rate (ESR) at 24 and longer weeks. | 12 week, 24week,36 week,48 week,72 week,96 week,120 week,144 week
  Change from baseline Erythrocyte Sedimentation Rate (ESR) at 24 and longer weeks.
Change from baseline C-Reactive Protein (CRP) at 24 and longer weeks. | 12 week, 24week,36 week,48 week,72 week,96 week,120 week,144 week
  Change from baseline C-Reactive Protein (CRP) at 24 and longer weeks.
Change from baseline swollen joint number (SW28) at 24 and longer weeks. | 12 week, 24week,36 week,48 week,72 week,96 week,120 week,144 week
  Change from baseline swollen joint number (SW28) at 24 and longer weeks. SW28 means the number of joints with swelling counted in 28 synovial joints, including proximal interphalangeal joints (10 joints), metacarpophalangeal joints (10), wrists (2), elbows (2), shoulders (2) and knees (2) bilateral.
Change from baseline tenderness joint number (T28) at 24 and longer weeks. | 12 week, 24week,36 week,48 week,72 week,96 week,120 week,144 week
  Change from baseline tenderness joint number (T28) at 24 and longer weeks. T28 means the number of joints with tenderness upon touching counted in 28 synovial joints, including proximal interphalangeal joints (10 joints), metacarpophalangeal joints (10), wrists (2), elbows (2), shoulders (2) and knees (2) bilateral.
Change from baseline patient global assessment(PGA) at 24 and longer weeks. | 12 week, 24week,36 week,48 week,72 week,96 week,120 week,144 week
  Change from baseline patient global assessment(PGA) at 24 and longer weeks.
Change from baseline physician global assessment(PHGA) at 24 and longer weeks. | 12 week, 24week,36 week,48 week,72 week,96 week,120 week,144 week
  Change from baseline physician global assessment(PHGA) at 24 and longer weeks.
Change from baseline Health Assessment Questionnaire (HAQ) at 24 and longer weeks. | 12 week, 24week,36 week,48 week,72 week,96 week,120 week,144 week
  Change from baseline Health Assessment Questionnaire (HAQ) at 24 and longer weeks.
Safety assessed by Adverse Events (AEs) | Up to 144 weeks
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product
Safety assessed by incidence of serious adverse events (SAE) | Up to 144 weeks
  Adverse Event is considered "serious" if the investigator or sponsor view any of the following outcomes: Death, life-threatening, persistent or significant disability/incapacity, congenital anomaly or birth defect, hospitalization, or medically important event.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Shu, Dr., Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data for all primary and secondary outcome measures will be made available within 12 months of study completion.